CLINICAL TRIAL: NCT01289691
Title: Atelectasis After Pulmonary Lobectomy: The Effect Of Air During One-Lung Ventilation (OLV) On Postoperative Atelectasis.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: London Health Sciences Centre (Other)
Responsible Party: Neal Badner, London Health Sciences Centre
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: LHSC2010AAPL
Record Dates: First submitted 2011-02-01; First posted 2011-02-04 (Estimated); Last update posted 2011-02-04 (Estimated); Status verified 2011-02

CONDITIONS: Pulmonary Atelectasis
Keywords: One Lung Ventilation; Atelectasis; Oxygenation
MeSH Terms: conditions — Pulmonary Atelectasis | interventions — One-Lung Ventilation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Air/Oxygen Mixture (Experimental): Patients in this group will be ventilated with a mixture of air and oxygen during one lung ventilation.
  Interventions: Other: One Lung Ventilation
- Oxygen (Active Comparator): Patients in this group will be ventilated with only oxygen during one lung ventilation.
  Interventions: Other: One Lung Ventilation

INTERVENTIONS:
Other: One Lung Ventilation — Patients in this group will be ventilated with a mixture of air and oxygen during one lung ventilation.
  Other Names: OLV
  Arms: Air/Oxygen Mixture
Other: One Lung Ventilation — Patients in this group will be ventilated with only oxygen during one lung ventilation.
  Other Names: OLV
  Arms: Oxygen

SUMMARY:
Patients scheduled for lung lobe resection using video assisted thoracic surgery will be randomly assigned to be ventilated with either only oxygen or a mixture of air and oxygen.

The primary purpose of this study is to determine if the incidence of postoperative collapse (in the non-surgical lung) is decreased when using a mixture of air and oxygen compared to using only oxygen (which is our control measurement) during one-lung ventilation.

DETAILED DESCRIPTION:
One of the concerns with all thoracic procedures employing One Lung Ventilation (OLV) is intra-operative hypoxia due to the large shunt that develops when only one lung is being ventilated. Ventilation with a higher fraction of inspired oxygen (FIO2) is one of the commonly chosen strategies for the treatment of hypoxemia during (OLV) for thoracic surgery. Using an FIO2 of 1.0 at all times during (OLV), however, may increase the risk of absorption atelectasis intra and postoperatively which itself leads to persistent hypoxia and potentially pneumonia.

The aim of this study is therefore to determine the impact of adding air to the inspired fraction of oxygen during (OLV) primarily on the incidence of postoperative atelectasis of the nonsurgical lung after lung resection using video assisted thoracic surgery and secondarily on intraoperative and postoperative oxygenation.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* Competent to give consent to enroll in study
* Booked for open thoracotomy procedure for lobectomy
* American Society of Anesthesiologists comorbidity score 1-4

Exclusion Criteria:

* Unable or unwilling to give consent
* Pregnant women
* Inability to insert an arterial line
* Severe COPD (FEV1 < .7% predicted, or FEV1/FVC < 0.70)
* Presence of other significant pulmonary impairment (PaO2 on room air 50 mmHg, PaCO2 > 50 mmHg or known pulmonary HTN mean PAP > 25 mmHg)
* Presence of significant cardiovascular disease (+MIBI that is non-revascularized, CCS ≥ 3 angina, NYHA ≥ 3 CHF, EF (by angiography or echocardiogram < 40%)
* Chronic renal failure (serum Cr > 200)
* Altered liver function

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2010-07; Primary Completion 2011-06 (Estimated); Study Completion 2011-06 (Estimated)

PRIMARY OUTCOMES:
The incidence of postoperative atelectasis | Immediately after the surgery - up to 2 days post operative.
  The primary objective is to determine if the incidence of postoperative atelectasis is decreased in the non-surgical lung, during one-lung ventilation (OLV) with mixture of air and oxygen compared to (OLV) using only oxygen (which is our control measurement) .

SECONDARY OUTCOMES:
The incidence of intraoperative and postoperative hypoxia (SpO2 < 90%) . | Intra-operative and Post operative day 1 and 2 .

CONTACTS AND LOCATIONS:
Overall Officials: Neal Badner, MD, FRCP(C), Principal Investigator — London Health Science Centre, University Of Western Ontario
Locations (1):
- Victoria Hospital, London, Ontario, Canada

REFERENCES:
- [Background] Rothen HU, Sporre B, Engberg G, Wegenius G, Hogman M, Hedenstierna G. Influence of gas composition on recurrence of atelectasis after a reexpansion maneuver during general anesthesia. Anesthesiology. 1995 Apr;82(4):832-42. doi: 10.1097/00000542-199504000-00004. PMID 7717553
- [Background] Schwarzkopf K, Klein U, Schreiber T, Preussetaler NP, Bloos F, Helfritsch H, Sauer F, Karzai W. Oxygenation during one-lung ventilation: the effects of inhaled nitric oxide and increasing levels of inspired fraction of oxygen. Anesth Analg. 2001 Apr;92(4):842-7. doi: 10.1097/00000539-200104000-00009. PMID 11273912
- [Background] Rothen HU, Sporre B, Engberg G, Wegenius G, Reber A, Hedenstierna G. Prevention of atelectasis during general anaesthesia. Lancet. 1995 Jun 3;345(8962):1387-91. doi: 10.1016/s0140-6736(95)92595-3. PMID 7760608